CLINICAL TRIAL: NCT04642495
Title: Clinical Application of Objective Visual Acuity Measurement Using Suppression Method to Inhibit Optokinetic Nystagmus (OKN).
Brief Title: Objective Visual Acuity Measurement Using Suppression of the Optokinetic Nystagmus (OKN).
Acronym: Speedwheel
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Anja Palmowski-Wolfe, Professor Dr. med., University of Basel
Other Study IDs: 2016-02078
Record Dates: First submitted 2020-11-17; First posted 2020-11-24 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Visual Acuity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Human subjects aged 4 and above: Human volunteers aged 4 and above.
  Interventions: Diagnostic Test: Visual acuity testing with SW , Landolt-"C" and Tumbling-"E" symbols

INTERVENTIONS:
Diagnostic Test: Visual acuity testing with SW , Landolt-"C" and Tumbling-"E" symbols — Establish prediction intervals for acuity tests

SUMMARY:
Suppression of the optokinetic nystagmus when a target is perceived can be applied to assess visual acuity objectively. Our aim is to establish prediction intervals for this optokinetic nystagmus suppression test (Speedwheel Test, SW) so that SW acuity may be used to estimate Snellen acuity (FrACT- C and -E) in the clinic in adults and children unable to cooperate in other acuity testing.

DETAILED DESCRIPTION:
In this prospective single center study subjects aged at least 4 years underwent testing of visual acuity with SW, Landolt-C and Tumbling-E symbols (Freiburg acuity test: FrACT-C, FrACT-E). Prediction intervals are to be established for SW compared to FrACT-C or -E and for FrACT- E compared to FrACT-C.

ELIGIBILITY:
Inclusion Criteria:

* able and willing to perform the test

Exclusion Criteria:

* under 4 years of age
* unable or unwilling

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy volunteers aged 4 and above
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Prediction intervals of Snellen acuity for the SW | 12 months
  Prediction intervals of Snellen acuity for the SW compared to Landolt C and E symbols

SECONDARY OUTCOMES:
Prediction intervals of Snellen acuity for Landolt C compared to E symbols | 12 months
  Prediction intervals of Snellen acuity for Landolt C compared to E symbols

CONTACTS AND LOCATIONS:
Overall Officials: Anja M Palmowski-Wolfe, Prof, Principal Investigator — University Basel, University Eye Hospital Basel
Locations (1):
- University Basel, University Eye Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
The results are to be shared in a publication

REFERENCES:
- [Background] Schwob N, Palmowski-Wolfe A. Objective measurement of visual acuity by optokinetic nystagmus suppression in children and adult patients. J AAPOS. 2019 Oct;23(5):272.e1-272.e6. doi: 10.1016/j.jaapos.2019.05.016. Epub 2019 Sep 14. PMID 31526857
- [Background] Schwob N, Palmowski-Wolfe A. Establishing an Objective Measurement of Visual Acuity with a Computerised Optokinetic Nystagmus Suppression Test. Klin Monbl Augenheilkd. 2020 Apr;237(4):502-505. doi: 10.1055/a-1119-6123. Epub 2020 Apr 24. PMID 32330979
- [Result] Luethy ML, Schotzau A, Palmowski-Wolfe A. Establishing Prediction Intervals for the SpeedWheel Acuity Test in Adults and Children. Klin Monbl Augenheilkd. 2021 Apr;238(4):488-492. doi: 10.1055/a-1403-2218. Epub 2021 Apr 14. PMID 33853189